CLINICAL TRIAL: NCT06085924
Title: Real World Evaluation of COVID-19 Burden and Nirmatrelvir/Ritonavir in Taiwan Using National Health Insurance Research Database
Brief Title: A Study to Learn About Effects of Living With COVID-19 and the Use of the Medicines Nirmatrelvir-Ritonavir in Treating COVID-19.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4671061; NCT06085924 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-10-16; First posted 2023-10-17 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: COVID-19
Keywords: COVID-19; real world evaluation on COVID-19 burden
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 - Cases of patients registered in the databases of all ages: Patients with a diagnosis of COVID-19 infection between 01 January 2021 and 31 December 2021
  Interventions: Other: Disease description
- Cohort 2 - Cases of patients registered in the databases of ≥12 years of age: Have COVID-19 diagnosis with international classification of diseases (ICD) code between 01 January 2022 and 31 December 2022
  Interventions: Drug: SoC

INTERVENTIONS:
Drug: SoC — COVID-19 treatment as per government guidance
  Groups: Cohort 2 - Cases of patients registered in the databases of ≥12 years of age
Other: Disease description — No intervention
  Groups: Cohort 1 - Cases of patients registered in the databases of all ages

SUMMARY:
The purpose of this study is to learn about:

* effects of living with COVID-19 and
* how effective is nirmatrelvir-ritonavir in treating COVID-19.

This is a study of two groups of COVID-19 patients in Taiwan.

In Group 1 the below participants were included in the study:

* Patients of all ages.
* Patients who were confirmed to have COVID-19 infection between 01 January 2021 and 31 December 2021.
* Cases of patients registered in the databases.

In Group 2 the below participants were included in the study:

* Participants who are 12 years or older.
* Confirmed to have COVID-19 between 01 January 2022 and 31 December 2022.

Nirmatrelvir-ritonavir is taken by mouth and is used to treat COVID-19.

The study will look at:

* the nature of Covid-19 disease.
* as well as the experiences of people receiving the nirmatrelvir-ritonavir.

This study will help to:

* understand what type of patients will need to be admitted to hospitals.
* see severe results due to COVID 19 infection.
* have more knowledge on the use of nirmatrelvir/ritonavir on COVID-19.

ELIGIBILITY:
Cohort 1:

Inclusion Criteria:

* Patients of all ages
* Patients with a diagnosis of COVID-19 infection between 01 January 2021 and 31 December 2021
* Cases of patients registered in the databases

Exclusion Criteria:

* Patients without COVID-19 diagnosis

Cohort 2:

Inclusion Criteria:

* ≥12 years of age
* Have COVID-19 diagnosis with international classification of diseases (ICD) code between 01 January 2022 and 31 December 2022

Exclusion Criteria:

* Patients without COVID-19 diagnosis

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study data will be retrospectively collected from the National Health Insurance Research Database (NHIRD). The NHIRD is a nation-wide claims database in Taiwan, which contains anonymized patient-level claims data covering 99.9% of the entire 23 million Taiwanese population.
Sampling Method: Non-Probability Sample
Enrollment: 8252912 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Cohort 1: Demographical Characteristics of Participants with a Diagnosis of COVID-19 That Required Intensive Care Unit (ICU) | 01 January 2021 to 31 December 2021
Cohort 1: Comorbidities of Participants with a Diagnosis of COVID-19 That Required ICU | 01 January 2021 to 31 December 2021
Cohort 1: Demographical Characteristics of Participants with a Diagnosis of COVID-19 That Did Not Require ICU | 01 January 2021 to 31 December 2021
Cohort 1: Comorbidities of Participants with a diagnosis of COVID-19 that did not require ICU | 01 January 2021 to 31 December 2021
Cohort 1: Demographical Characteristics of Participants with a diagnosis of COVID-19 that required ICU | 01 January 2021 to 31 December 2021
Cohort 1: Demographical Characteristics of Participants with a Diagnosis of COVID-19 That Required Ventillatory Support | 01 January 2021 to 31 December 2021
Cohort 1: Comorbidities of Participants with a Diagnosis of COVID-19 That Required Ventillatory Support | 01 January 2021 to 31 December 2021
Cohort 1: Demographical Characteristics of Participants with a Diagnosis of COVID-19 That Did Not Require Ventillatory Support | 01 January 2021 to 31 December 2021
Cohort 1: Comorbidities of Participants with a Diagnosis of COVID-19 That Did Not Require Ventillatory Support | 01 January 2021 to 31 December 2021
Cohort 1: Demographics of Participants with a Diagnosis of COVID-19 That Had a Fatal Outcome | 01 January 2021 to 31 December 2021
Cohort 1: Comorbidities of Participants with a Diagnosis of COVID-19 That Had a Fatal Outcome | 01 January 2021 to 31 December 2021
Cohort 1: Demographics of Participants with a Diagnosis of COVID-19 That Did Not Have a Fatal Outcome | 01 January 2021 to 31 December 2021
Cohort 1: Comorbidities of Participants with a Diagnosis of COVID-19 That Did Not Have a Fatal Outcome | 01 January 2021 to 31 December 2021
Cohort 2: Characteristics Associated with Patients Receiving nirmatrelvir/ritonavir vs Patients Not Receiving nirmatrelvir/ritonavir | 01 January 2022 to 31 December 2022

SECONDARY OUTCOMES:
Cohort 1: Demographics of Participants with a Diagnosis of COVID-19 That Required Hospital Admission | 01 January 2021 to 31 December 2021
Cohort 1: Comorbidities of Participants with a Diagnosis of COVID-19 That Required Hospital Admission | 01 January 2021 to 31 December 2021
Cohort 1: Demographics of Participants with a Diagnosis of COVID-19 That Did Not Require Hospital Admission | 01 January 2021 to 31 December 2021
Cohort 1: Comorbidities of Participants with a Diagnosis of COVID-19 That Did Not Require Hospital Admission | 01 January 2021 to 31 December 2021
Cohort 1: Incidence Proportion of ICU Admissions Among COVID-19 Patients Requiring Hospitalization Per Age Range | 01 January 2021 to 31 December 2021
Cohort 1: Clinical Characteristics Associated to ICU Admission Among Hospitalized COVID-19 Patients | 01 January 2021 to 31 December 2021
Cohort 1: Risk Factors Associated to ICU Admission Among Hospitalized COVID-19 Patients | 01 January 2021 to 31 December 2021
Cohort 1: Clinical Characteristics Associated to Ventilatory Support Among Hospitalized COVID-19 Patients | 01 January 2021 to 31 December 2021
Cohort 1: Risk Factors Associated to Ventilatory Support Among Hospitalized COVID-19 Patients | 01 January 2021 to 31 December 2021
Cohort 1: Mortality Rate Associated to Ventilatory Support Among Hospitalized COVID-19 Patients | 01 January 2021 to 31 December 2021
Cohort 1: Average Length of Stay (LOS) of Hospitalized COVID-19 Patients | 01 January 2021 to 31 December 2021
Cohort 2: Incidence for severe COVID-19 Overall | 01 January 2022 to 31 December 2022
Cohort 2: Incidence for severe COVID-19 By Risk Group | 01 January 2022 to 31 December 2022
Cohort 2: Incidence for severe COVID-19 By Time Period | 01 January 2022 to 31 December 2022
Cohort 2: Relative Risk for severe COVID-19 Overall | 01 January 2022 to 31 December 2022
Cohort 2: Relative Risk for severe COVID-19 By Risk Group | 01 January 2022 to 31 December 2022
Cohort 2: Relative Risk for severe COVID-19 By Time Period | 01 January 2022 to 31 December 2022

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Taiwan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671061